CLINICAL TRIAL: NCT04527497
Title: Clinical Course and Treatment of COVID-19 Inpatients in Hospital
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Other Study IDs: WI_20-1294
Record Dates: First submitted 2020-08-20; First posted 2020-08-26 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is an epidemiological observational study. It serves to collect data from patients with positive COVID-19 test results who are hospitalized. All data describing the course of the inpatient stay are recorded (Length of stay, course of therapy, medication, X-ray and CT results,ventilation mode and duration, laboratory). Furthermore, anthropometric data and information on COVID-19 symptoms is recorded.

DETAILED DESCRIPTION:
The aim of this study is to describe the course of disease and the treatment of patients suffering from COVID-19 who are hospitalized and treated as inpatients:

1. Are there common features (previous illnesses, medication, age, BMI, etc.), which may influence the course of disease?
2. Are there therapeutic procedures that have a positive or negative impact on the course of the disease or the length of stay in the intensive care unit/ the duration of ventilation (early/late intubation, CPAP, NIV, ECMO)?

ELIGIBILITY:
Inclusion Criteria:

* positive COVID-19 test result
* Age > 18 years

Exclusion Criteria:

* Age < 18 years
* negative COVID-19 test result
* lack of agreement
* Any medical, psychological or other condition, that restricts the ability of the person to be informed and to give the consent for voluntary participation in this trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who are inpatients at Bethanien Hospital and have a proven COVID-19 infection and who agree to participate in the study during the period from 01.08.2020 - 30.05.2021.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
convalescence/death | through study completion, an average of 2 months
  has patient died or has patient recovered

SECONDARY OUTCOMES:
length of stay in the intensive care unit | through study completion, an average of 2 months
  length of stay in the intensive care unit
length of stay in hospital | through study completion, an average of 2 months
  length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Randerath, Prof. Dr., Principal Investigator — Krankenhaus Bethanien Solingen
Locations (1):
- Institut für Pneumologie an der Universität zu Köln / Wissenschaftliches Institut Bethanien für Pneumologie e.V., Solingen, North Rhine-Westphalia, Germany